CLINICAL TRIAL: NCT02742740
Title: Embodied Conversational Agent (ECA) as an Oncology Trial Advisor
Brief Title: Study Buddy (an ECA Oncology Trial Advisor) for Cancer Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Northeastern University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael Paasche-Orlow, Associate Professor, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-34989; 5R01CA158219-05 (NIH)
Record Dates: First submitted 2016-04-06; First posted 2016-04-19 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Patient Satisfaction; Patient Compliance; Guideline Adherence
MeSH Terms: conditions — Patient Satisfaction; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard of care for chemotherapy treatment.
- Chemo Buddy (Experimental): Subject receives instructions on how to use the personalized touch screen tablet and takes it home for 2 months.
  Interventions: Behavioral: Chemo Buddy

INTERVENTIONS:
Behavioral: Chemo Buddy — The Study Buddy ECA acts as an advisor to patients on chemotherapy regimens, promoting protocol adherence and retention, providing anticipatory guidance and answering questions, serving as a conduit to capture information about complaints or adverse events, providing a venue for communicating about updates.
  Arms: Chemo Buddy

SUMMARY:
The Study Buddy ECA acts as an advisor to patients on chemotherapy regimens, promoting protocol adherence and retention, providing anticipatory guidance and answering questions, serving as a conduit to capture information about complaints or adverse events, providing a venue for communicating about updates. The Study Buddy will use the web-based ECA infrastructure developed for use on another project. We will use web browsers on tablets provided to study participants to access the Study Buddy, providing anywhere, anytime access to its functions. Usability metrics will include session time, satisfaction, and error rates.

DETAILED DESCRIPTION:
Subjects will be identified from among patients on chemotherapy regimens at BMC. With the provider's approval, we will recruit patients for this study.

All subjects will be enrolled for 2 months. After consent, we will collect baseline data. Baseline data is collected after enrollment and before randomization. Baseline data includes:

sociodemographic data PROMIS Mental and Social health the PHQ-9 clinical factors such as medical diagnosis (cancer type and stage) the Short Assessment of Health Literacy-English the Short Portable Mental Status Questionnaire (SPMSQ) for cognitive impairment the Need For Cognition scale contact numbers of two friends or family members who will assist us in establishing contact, if necessary.

The exit interview will be conducted 2 months after the baseline interview, with windows of 2 weeks plus or minus that date. Study staff will attempt to coincide this interview with a clinical visit, to minimize inconvenience for the subject.

Data collected at the exit interview will include:

PROMIS Mental and Social health the PHQ-9 Satisfaction with ECA

Review of the subject's medical chart will be performed bi-weekly while the subject is enrolled. Chart review will be performed by a staff member who is blinded to the subject's group (intervention vs control).

ELIGIBILITY:
Inclusion Criteria:

1. speaks English fluently
2. is able to independently consent into this study and parent cancer study
3. has adequate corrected vision to use the ECA system (based on a 1-minute functional screener)
4. has adequate hearing to use the ECA system

Exclusion Criteria:

1. suicidal or homicidal
2. currently in police custody
3. do not live in the Boston area
4. plan on leaving the Boston area for more than 4 weeks in the next 6 months
5. score 6 or less on the SPMSQ screening test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
treatment protocol adherence | up to 8 weeks
  How well does the subject adhere to treatment protocol. This will be defined by the number of treatment visits attended/ number of treatment visits scheduled [excluding any treatment visits that have been cancelled by the clinicians].

SECONDARY OUTCOMES:
Subject Satisfaction | assessed at 2 months
  assessed by questionnaire
Number of adverse events | assessed at 2 months
  as reported through tablet and directly to clinic by patient
time to detect and resolve adverse events | assessed at 2 months
  as reported through tablet and directly to clinic by patient
adverse event false alarm rate | assessed at 2 months
  as reported through tablet and directly to clinic by patient

CONTACTS AND LOCATIONS:
Overall Officials: Michael Paasche-Orlow, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No